# **Study Protocol**

Title: Multigene Panel Test in Gastric Cancer Patients in Portugal

NCT:

Date: 01 September 2024.

#### **Authors:**

- 1. Mourato B., MD
  - a. Affiliation: Unidade Local de Saúde do Norte Aletenjano;
  - b. Contacts: email: <u>beatriz.mourato@ulsna.min-saude.pt</u>; Address: Hospital Doutor José
     Maria Grande, Avenida de Santo António, 7300-853, Portalegre;
  - c. Contributions: Main author; Study designer.
- 2. Areia M., PhD
  - a. Affiliation
    - i. Instituto Português de Oncologia de Coimbra;
    - ii. RISE@CI-IPO (Health Research Network), Portuguese Oncology Institute of Porto (IPO Porto)
  - b. Contacts: email: miguel.areia75@gmail.com; Address: Avenida Bissaya Barreto 98, 3000-075 Coimbra.
  - c. Contributions: Intellectual contributor; Reviewer.
- 3. Fronteira, I., PhD
  - a. Affiliation:
  - b. Contacts: ines.fronteira@ensp.unl.pt; Address: Avenida Padre Cruz, 1600-560 Lisboa.
  - c. Contributions: Study designer; Intellectual contributor; Reviewer.
- 4. Dinis, R., PhD
  - a. Affiliation: Hospital do Espírito Santo de Évora,
  - b. Contacts: email: <u>rui.p.dinis@ulsna.min-saude.pt</u>; Address: Largo do Sr. Da Probreza, 7000-811 Évora;
  - c. Contributions: Study designer; Study collaborator; Reviewer.

#### **Abstract**

Abstract: Gastric cancer (GC) is the fifth with the highest incidence and mortality worldwide (1). It is a multifactorial and heterogeneous disease, where both environmental and genetic factors are involved. Three hereditary syndromes primarily affect the stomach: Hereditary Diffuse Gastric Cancer (HDGC), Gastric Adenocarcinoma and Stomach Proximal Polyposis (GAPPS), and Familial Intestinal Gastric Cancer (FIGC) (2), but in addition to these, many other syndromes and genetic mutations are associated with an increased risk of GC (3–5). As GC is a neoplasm with numerous somatic and hereditary mutations involved in its carcinogenesis, the use of the Multigene Germline Panel Test (MGPT) may be crucial, as it allows the analysis of hereditary mutations in a significant number of genes simultaneously (6,7). This observational, retrospective study aims to quantify and characterise the pathogenic variants (PVs) found in the MGPT of GC patients in Alto Alentejo (Portugal).

#### Introduction

# Background/ Rationale

According to data from the Global Cancer Observatory, gastric cancer (GC) ranks fifth in terms of incidence and mortality worldwide (1).

It is a multifactorial and heterogeneous disease involving both environmental and genetic factors. Although the majority of cases are sporadic, caused by environmental exposures, up to 20% of patients have a familial aggregation and of these, 3 to 5% are classified as hereditary with an identified mutation (8,9). Three hereditary syndromes primarily affect the stomach: Hereditary Diffuse Gastric Cancer (HDGC); Gastric Adenocarcinoma and Stomach Proximal Polyposis (GAPPS); and Familial Intestinal Gastric Cancer (FIGC) (2). HDGC is an autosomal dominant syndrome, predominantly caused by germline mutations in the CDH1 gene, which encodes the e-cadherin protein with important functions in cell aggregation, and is characterised by a high risk of early-onset diffuse GC and invasive lobular breast cancer (10). GAPPS is caused by germline mutations in APC promoter 1B and is characterised by the presence of fundic gland polyposis with focal dysplasia and intestinal or mixed adenocarcinoma at the level of the gastric fundus and sparing the antrum (4,11). Finally, FIGC is an autosomal dominant syndrome, still poorly characterized genetically, which is associated with an increased risk of intestinal GC (10).

Other genetic syndromes are also associated with an increased risk of GC. Some of the genes involved include MLH1, MSH2, MSH6, and PMS2 (Lynch Syndrome - LS), TP53 (Li-Fraumeni Syndrome), APC (PAF and ADC / proximal polyposis of the stomach) and MUTYH (Polyposis Associated MUTYH), BMPR1A and SMAD4 (Juvenile Polyposis Syndrome), STK11 (Peutz-Jegher Syndrome) and PTEN (Cowden Syndrome) (3–5).

As GC is a neoplasm with numerous somatic and hereditary mutations involved in its carcinogenesis, the use of MGPT can be crucial, as it performs the analysis of hereditary mutations in a significant number of genes simultaneously (depending on the genes included in the panel) (6,7). In addition to the described mutations, MGPT has allowed the identification of new genetic mutations associated with GC risk, including in the BRCA 1/2, PALB2, ATM and RAD51C genes (typically associated with hereditary breast and ovarian cancer), MAP3K6,

MYD88, among others (9,12–17). However, the use of MGPT, especially in unselected GC patients, is not without risks, such as the unexpected detection of PV in genes not strictly associated with the phenotype (secondary findings) or, more commonly, the high rate of variants of unknown significance (VUS), which can raise important questions regarding the uncertainty of how to approach these patients (18). Therefore, some studies advocate that MGPT or single gene testing (SGT) should be offered only to selected patients, especially those with suspected HDCG (5,19–21). On the other hand, the evidence of many other germline mutations associated with GC and the lack of genetic characterisation of FIGC justifies the growing interest in performing MGPT in unselected patients with GC (10,18,22,23). Although these studies suggest abenefit in the use of MGPT in unselected patients with GC, this test is not yet widely used.

In Portugal, the incidence and mortality rates of GC have been increasing over the last few decades. It is therefore important to better understand the genetic characteristics of GC in this country in order to develop better strategies for managing this disease.

# **Objectives**

The **main objective** of this research is to quantify and characterize the PV found in MGPT of GC patients in Alto Alentejo (Portugal).

## The **specific objectives** are:

- Determine the global rate of PVs in GC patients of Alto Alentejo;
- Determine which PVs are most common in our GC population;
- Correlate the PVs found with clinical factors: Age at diagnosis; Sex; Weight; Height; Presence of other diseases (Diabetes; Arterial Hypertension; Dyslipidaemia; Stroke; Heart attack); Date of diagnosis; Stage at diagnosis; Histologic subtype; Surgery for GC; Personal history of other cancers; Familial history of GC and other cancers;
- Correlate the PVs found with prognostic factors: 12-month survival rate; mortality.

#### Methods

#### Study design

Observational, retrospective study

Despite this design, there was uniformity in the data recorded for each participant who agreed to be submitted to MGPT, minimizing the variability between records or the missing clinical data.

## **Setting**

This study takes place at the Unidade Local de Saúde do Alto Alentejo (ULSAALE). The MGPT was always performed in the same laboratory (Germano de Sousa – Centro de Genética Laboratorial) using peripheral blood samples from patients with GC.

Two types of MGPT were used:

- MGPT 4005 (15 genes): APC, ATM, BLM, BMPR1A, CDH1, CTNNA1, EPCAM, MLH1, MSH2, MSH6, PMS2, PTEN, SMAD4, STK11TP53.
- MGPT 4013 (30 genes): ATM, BARD1, BLM, BRCA1, BRCA2, BRIP1, CDH1, CHEK2, EPCAM, FANCC, MLH1, MRE11A, MSH2, MSH6, MUTYH,

NBN, NF1, PALB2, PMS2, PTEN, RAD50, RAD51C, RAD51D, RECQL4, RINT1, SLX4, SMARCA4, STK11, TP53, XRCC2.

The majority of patients with GC were tested with MGPT 4005. Patients with neoplasms other than GC or with a family history of other neoplasms were tested with MGPT 4013. The decision to perform MGPT and the choice of panel type were made in multidisciplinary consultation.

The recruitment process takes place between January 2023 and December 2024. All data will be collected and entered in a database until September 2025

The manuscript for publication will be written between October and November 2025.

# **Participants**

Eligibility criteria:

- Adult patients (over 18 years old) with a histologically proven diagnosis
  of gastric adenocarcinoma that have done MGPT between 2023 and
  2024;
- Ability to understand and speak Portuguese and/or English language;
- Ability to reliably provide informed consent for inclusion in the study.

There are no matched or randomized groups.

# Variables / Measurement

Table 2

#### **Data sources**

The variables related to the patient's clinical history and personal data will be collected through a questionnaire administered during a personal interview and supplemented by consultation of each patient's digital medical record in order to obtain more detailed information on the variables characterising the disease and the results of the MGPT.

## Bias

Efforts to address potential sources of bias:

Clear Inclusion and Exclusion Criteria: The inclusion criteria are clear to select patients that are representative of the target population (patients with gastric adenocarcinoma) and that there is no bias in participant selection.

Control of Confounding Factors: There are some confounding factors that may influence the study results, such as age, sex, Weight; Height; Body mass index; Presence of other diseases: Diabetes; Arterial Hypertension; Dyslipidaemia; Stroke; Heart attack). This will be achieved through appropriate statistical techniques or data stratification during analysis.

Uniformity in data records: There was uniformity in the data recorded for each participant who agreed to be submitted to MGPT, minimizing the variability between records or the missing clinical data.

Consistent and Accurate Data Collection: This will be achieved through adequate training of interviewers or data collection personnel and the use of standardized data collection protocols.

Blind Data Assessment: After collection, the data will be pseudo-anonymized so that the researcher who analyses the data will not have access to the patient's identifying data.

Time-Sensitive Analysis: Data analysis takes into account the timing of data collection relative to relevant clinical events.

Sensitivity Analysis: It will be performed a sensitivity analyses to assess the robustness of the results across different results of MGPT and clinical factors.

## Study size

The sample calculation takes into account the number of annual cases of GC recorded in Alto Alentejo (65 cases in 2020, data from National Oncologic Registry). Therefore, the sample calculation suggests that it should include 56 patients with GC, with a confidence level of 95% and a margin of error of 5%.

# Quantitative variables

For quantitative variables we will do the descriptive statistics analyses with mean, mode, median, standard deviation, interquartile variation, maximum and minimum.

Subgroup analysis will be carried out, for each quantitative and qualitative variable, dividing patients who have positive or negative MGPT. We will analyse the effect measures of the difference between the two groups, with confidence interval (IC) 95%, and if possible, inferential statistical analysis will be conducted.

# Statistical methods

- a) Statistical analysis will be carried out using SPSS software.
- b) In inferential statistical analysis, the normality of the distribution of quantitative variables will be determined by the Kolmogorov-Smironov test. For variables with normal distribution, the T-sudent test will be used and for those that do not have normal distribution, the Mann-Whitney test will be performed, with the purpose of analysing the statistical significance of the difference between the groups with IC 95% (positive MGPT and negative MGPT). For qualitative variables, the statistical significance of the difference between groups, with 95% CI, will be calculated using the Chi-square test (if more than 10% of the cells in the 2x2 tables have frequencies ≤5) or the Exact Fisher Test. We will later perform a multivariate analysis with logistic regression to control confounding variables.
- c) Missing data: We addressed missing data by employing multiple strategies. Firstly, we conducted a thorough examination of patterns of missingness to discern if they followed a missing completely at random, missing at random, or missing not at random pattern. Subsequently, for cases with missing data, we utilized multiple imputation techniques to impute missing values based on observed data and variables that were predictive of missingness. Additionally, we performed sensitivity analyses to assess the robustness of our findings to different assumptions regarding the missing data mechanism. Overall, these

- approaches allowed us to minimize bias and maintain the integrity of our analyses in the presence of missing data.
- d) To conduct sensitivity analysis for this study, we will systematically vary key parameters or assumptions within our analytical framework to assess their impact on the study outcomes. This may involve testing different statistical models, criteria for participant inclusion/exclusion, handling of missing data, or adjustments for potential confounding variables. By exploring a range of scenarios, we aim to evaluate the robustness of our findings and assess the degree to which they are influenced by specific methodological choices or assumptions. Sensitivity analysis allows us to identify the potential sources of uncertainty and to provide a more comprehensive understanding of the reliability and generalizability of our study results.

**Table 2 - Variables / Measurements** 

| Type of Variable | Name of Variable | Measurements |
|---|---|---|
| MGPT Outcomes<br>variables | MGPT | positive (1) or negative (0) |
| | PV | integer number |
| | Likely pathogenic variables (LP) | integer number |
| | Name of genes with PV | descriptive |
| | PV in each gene | integer number |
| | vus | integer number |
| Potential<br>confounders<br>variables | Age at diagnosis | Years |
| | Sex | Female(1)/Male(0) |
| | Weight | Kg |
| | Height | cm |
| | Body mass index | Kg/m <sup>2</sup> |

| | Presence of other diseases: Diabetes; Arterial Hypertension; Dyslipidaemia; Stroke; Heart attack); | Yes(1)/No(0) for each disease |
|---|---|---|
| | Stage at diagnosis (AJCC staging system); | 0, I, IIa, IIb, III, IVa, IVb |
| | Histologic subtype; | Intestinal (1); Diffuse (2); Mixed (3) |
| "Exposures"<br>variables | Personal history of other cancers | Yes (1)/No (0) |
| | Types of other cancer in GC patient | descriptive |
| | Familial history of GC | Yes (1)/No (0) |
| | Age of onset of each familial case of GC | integer number |
| | Familial history of other cancers (specifying) | descriptive |
| | Age of onset of each familial case of other cancers | Years |
| Prognostic<br>related variables | 12-months survival | Yes (1)/No(0) |
| | Death due to GC | Yes (1)/No(0) |
| | Date of death | mm/yyyy |
| Other variables: | Date of diagnosis | mm/yyyy |
| | Localization of tumor | Cardia / Fundos / Body / Antrum/pyloro |
| | Time since diagnosis until the current moment | months |
| | Surgery for GC | Yes (1)/No (0); |
| | Type of surgery | Total gastrectomy (1); Subtotal gastrectomy (0) |
| | Date of Surgery | mm/yyyy |
| | Histologic staging after surgery | 0, I, IIa, IIb, III, IVa, IVb |
| | Underwent chemotherapy | Yes (1) / No (0) |
| | Type of chemotherapy | descriptive |

| Cycles of chemotherapy | integer number |
|------------------------|----------------|

Positive MGPT is considered when it is found at least one PV in one gene of teste

A comparative analysis will be made between the individual characteristics and tumor characteristics of positive MGPT cases with those with negative MGPT.

#### **Ethical Issues**

This research has already been approved by the Ethics Committee and the Board of Directors of ULSAALE (Ata 06/2024, document 60 / 202400991) and it will be submitted to Ethics Committee of the Nova Medical School.

Participation in the study is voluntary, with informed consent and participants will be informed of the results before publication.

# **Risks and Benefits**

The main benefits and expected outcomes of the study are the contribution to a better understanding of GC carcinogenesis, which could improve the diagnostic and therapeutic approach of GC patients and their relatives. In addition, this research may help to clarify whether the prevalence of hereditary GC is higher than that described in the literature (3-5%) (4,5), and may justify screening the population for this disease.

However, the use of MGPT is not without important risks, namely the identification of variants of undetermined significance (VUS), which requires careful integration of all clinical and genetic information for correct personal and family counselling. Whenever necessary, VUS carriers (as well as patients with identified PVs) will be referred to the Portuguese Institute of Oncology in Lisbon (IPOLFG) for family risk and genetic counselling. Other potential risks of this study include the psychological stress and anxiety caused by the survey and MGPT results, the need to travel to participate in the study, and the fact that the study is being conducted by non-geneticist researchers, which limits the immediate counselling that can be provided. In this way, we will have the collaboration of the psychologists of the Day Hospital, and our close collaboration with the Germano de Sousa Genetics Laboratory and the IPOLFG teams will allow an adequate response to technical questions about the MGPT. Finally, it should be noted that this observational study will only analyse the MGPT results of CG patients and will not propose any additional intervention for patients or their families.

#### References

- 1. International Agency for Research on Cancer. Global Cancer Observatory 2022 Stomach. 2022.
- 2. Gullo I, Van Der Post RS, Carneiro F. Recent advances in the pathology of heritable gastric cancer syndromes. Histopathology. 2021 Jan;78(1):125–47.
- 3. Van Der Post RS, Vogelaar IP, Carneiro F, Guilford P, Huntsman D, Hoogerbrugge N, et al. Hereditary diffuse gastric cancer: updated clinical guidelines with an emphasis on germline *CDH1* mutation carriers. J Med Genet. 2015 Jun;52(6):361–74.
- 4. Li J, Woods SL, Healey S, Beesley J, Chen X, Lee JS, et al. Point Mutations in Exon 1B of APC Reveal Gastric Adenocarcinoma and Proximal Polyposis of the Stomach as a Familial Adenomatous Polyposis Variant. Am J Hum Genet. 2016 May;98(5):830–42.
- 5. Tedaldi G, Pirini F, Tebaldi M, Zampiga V, Cangini I, Danesi R, et al. Multigene Panel Testing Increases the Number of Loci Associated with Gastric Cancer Predisposition. Cancers. 2019 Sep 11;11(9):1340.
- 6. Yurgelun MB, Allen B, Kaldate RR, Bowles KR, Judkins T, Kaushik P, et al. Identification of a Variety of Mutations in Cancer Predisposition Genes in Patients With Suspected Lynch Syndrome. Gastroenterology. 2015 Sep;149(3):604-613.e20.
- 7. Dahui Q. Next-generation sequencing and its clinical application. Cancer Biol Med. 2019 Feb 1;16(1):4–10.
- 8. Machlowska J, Baj J, Sitarz M, Maciejewski R, Sitarz R. Gastric Cancer: Epidemiology, Risk Factors, Classification, Genomic Characteristics and Treatment Strategies. Int J Mol Sci. 2020 Jun 4;21(11):4012.
- 9. Hansford S, Kaurah P, Li-Chang H, Woo M, Senz J, Pinheiro H, et al. Hereditary Diffuse Gastric Cancer Syndrome: *CDH1* Mutations and Beyond. JAMA Oncol. 2015 Apr 1;1(1):23.
- 10.Carneiro F. Familial and hereditary gastric cancer, an overview. Best Pract Res Clin Gastroenterol. 2022 Jun;58–59:101800.
- 11.Worthley DL, Phillips KD, Wayte N, Schrader KA, Healey S, Kaurah P, et al. Gastric adenocarcinoma and proximal polyposis of the stomach (GAPPS): a new autosomal dominant syndrome. Gut. 2012 May;61(5):774–9.
- 12. Majewski IJ, Kluijt I, Cats A, Scerri TS, De Jong D, Kluin RJ, et al. An  $\alpha$ -E-catenin ( *CTNNA1* ) mutation in hereditary diffuse gastric cancer. J Pathol. 2013 Mar;229(4):621–9.
- 13. Gaston D, Hansford S, Oliveira C, Nightingale M, Pinheiro H, Macgillivray C, et al. Germline Mutations in MAP3K6 Are Associated with Familial Gastric Cancer. Horwitz MS, editor. PLoS Genet. 2014 Oct 23;10(10):e1004669.
- 14. Fewings E, Larionov A, Redman J, Goldgraben MA, Scarth J, Richardson S, et al. Germline pathogenic variants in PALB2 and other cancer-predisposing genes in families with hereditary diffuse gastric

- cancer without CDH1 mutation: a whole-exome sequencing study. Lancet Gastroenterol Hepatol. 2018 Jul;3(7):489–98.
- 15. Vogelaar IP, Van Der Post RS, Van Krieken JHJ, Spruijt L, Van Zelst-Stams WA, Kets CM, et al. Unraveling genetic predisposition to familial or early onset gastric cancer using germline whole-exome sequencing. Eur J Hum Genet. 2017 Nov;25(11):1246–52.
- 16.Weren RDA, Van Der Post RS, Vogelaar IP, Van Krieken JH, Spruijt L, Lubinski J, et al. Role of germline aberrations affecting *CTNNA1*, *MAP3K6* and *MYD88* in gastric cancer susceptibility. J Med Genet. 2018 Oct;55(10):669–74.
- 17. Slavin T, Neuhausen SL, Rybak C, Solomon I, Nehoray B, Blazer K, et al. Genetic Gastric Cancer Susceptibility in the International Clinical Cancer Genomics Community Research Network. Cancer Genet. 2017 Oct;216–217:111–9.
- 18.Calvello M, Marabelli M, Gandini S, Marino E, Bernard L, Dal Molin M, et al. Hereditary Gastric Cancer: Single-Gene or Multigene Panel Testing? A Mono-Institutional Experience. Genes. 2023 May 13;14(5):1077.
- 19. Carvalho J, Oliveira P, Senz J, São José C, Hansford S, Teles SP, et al. Redefinition of familial intestinal gastric cancer: clinical and genetic perspectives. J Med Genet. 2021 Jan;58(1):1–11.
- 20.Hossain MU, Ahammad I, Moniruzzaman Md, Akter Lubna M, Bhattacharjee A, Mahmud Chowdhury Z, et al. Investigation of pathogenic germline variants in gastric cancer and development of "GASCANBASE" database. Cancer Rep. 2023 Dec;6(12):e1906.
- 21. Aronson M, Swallow C, Govindarajan A, Semotiuk K, Cohen Z, Kaurah P, et al. Germline Variants and Phenotypic Spectrum in a Canadian Cohort of Individuals with Diffuse Gastric Cancer. Curr Oncol. 2020 May 1;27(2):182–90.
- 22.Uson PLS, Kunze KL, Golafshar MA, Botrus G, Riegert-Johnson D, Boardman L, et al. Germline Cancer Testing in Unselected Patients with Gastric and Esophageal Cancers: A Multi-center Prospective Study. Dig Dis Sci. 2022 Nov;67(11):5107–15.
- 23. Bilyalov A, Nikolaev S, Danishevich A, Khatkov I, Makhmudov K, Isakova Z, et al. The Spectrum of Germline Nucleotide Variants in Gastric Cancer Patients in the Kyrgyz Republic. Curr Issues Mol Biol. 2023 Jul 31;45(8):6383–94.